CLINICAL TRIAL: NCT03769233
Title: A 5-week Mindfulness Program for Emerging Adults Experiencing Anxious and/or Depressive Symptoms
Brief Title: Mindfulness for Emerging Adults Experiencing Anxious and/or Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Dr. Jennine Rawana, Associate Professor & Clinical Developmental Psychologist, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2018-349
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Depressive Symptoms; Anxious Symptoms
Keywords: Mindfulness; Well-being; Emotion Regulation; Perceived Stress; Self-Compassion
MeSH Terms: conditions — Depression; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based Intervention (Experimental): 5 week, manual-based group MBI treatment for depressive and anxious symptoms
  Interventions: Behavioral: Mindfulness-based Intervention

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention — MBI will be delivered in group format, 90 minutes per week, for 5 consecutive weeks with 6-15 participants per group.

SUMMARY:
Emerging adults (EA; 18 to 29 years old) in Canada are among the age group with highest risk of developing mental health issues. Despite this, they experience especially long wait-times for mental health services. To date, there has been minimal research into developmentally appropriate treatment options for the EA population. Mindfulness-based interventions (MBIs) are emerging as a potential treatment to address this need. MBIs are group-based psychological treatments for coping with distress, with the goal of improving mental health. Unfortunately, these 'traditional' MBIs are very demanding in terms of time and homework and are therefore not sufficiently feasible for the demanding schedules of EA university students. Instead, recent studies suggest a role for briefer MBIs in addressing mental health symptom burden, well-being and reducing acute stress symptoms. The brevity of these interventions make them theoretically better suited for EA university populations. High quality research, including controlled clinical trials are needed to demonstrate whether MBIs can provide efficacious treatment to improve the lives of EA university students. The current study will test the efficacy of a five-week MBI baseline within-subject controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* consenting Emerging Adults
* Ability to communicate, in written and spoken English

Exclusion Criteria:

* Minimal depressive and anxious symptoms (score below 10 and 8 on the PHQ-9/GAD-7
* Current substance abuse or dependence, psychosis or mania
* Current self-injurious behavior of past suicide attempt
* Previously completed >4 weeks of an MBI, or general Cognitive behavioral Therapy, in the past 3 years

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Depressive Symptoms at 2.5 Weeks, 5 Weeks, 7.5 Weeks and 11.5 Weeks | Baseline (Week 0), Pre- (Week 2.5), Mid- (Week 5), Post-Treatment (Week 7.5), and 1-month Follow-up (Week 11.5
  Patient Health Questionnaire-9 (PHQ-9): Scale used to measure Depressive Symptoms, with higher scores reflecting greater levels of depressive symptoms
Change from Baseline Anxious Symptoms at 2.5 Weeks, 5 Weeks, 7.5 Weeks and 11.5 Weeks | Baseline (Week 0), Pre- (Week 2.5), Mid- (Week 5), Post-Treatment (Week 7.5), and 1-month Follow-up (Week 11.5)
  Generalized Anxiety Disorder-7 (GAD-7): Scale used to measure Anxious Symptoms, with higher scores reflecting greater levels of anxious symptoms
Change from Baseline Mental Wellbeing at 2.5 Weeks, 5 Weeks, 7.5 Weeks and 11.5 Weeks | Baseline (Week 0), Pre- (Week 2.5), Mid- (Week 5), Post-Treatment (Week 7.5), and 1-month Follow-up (Week 11.5)
  Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS): Scale used to measure Mental Wellbeing, with higher scores reflecting greater levels of mental wellbeing

SECONDARY OUTCOMES:
Change from Baseline Perceived Stress at 2.5 Weeks, 5 Weeks, 7.5 Weeks and 11.5 | Baseline (Week 0), Pre- (Week 2.5), Mid- (Week 5), Post-Treatment (Week 7.5), and 1-month Follow-up (Week 11.5)
  10-item Perceived Stress Scale (PSS-10): Scale used to measure Perceived Stress, with higher scores reflecting greater levels of perceived stress
Change from Baseline Emotion Regulation Strategies at 2.5 Weeks, 5 Weeks, 7.5 Weeks and 11.5 | Baseline (Week 0), Pre- (Week 2.5), Mid- (Week 5), Post-Treatment (Week 7.5), and 1-month Follow-up (Week 11.5)
  Emotion Regulation Questionnaire (ERQ): Scale used to measure Emotion Regulation, with higher scores reflecting greater levels of emotion regulation strategies
Change from Baseline Self-Compassion at 2.5 Weeks, 5 Weeks, 7.5 Weeks and 11.5 | Baseline (Week 0), Pre- (Week 2.5), Mid- (Week 5), Post-Treatment (Week 7.5), and 1-month Follow-up (Week 11.5)
  Self-Compassion Scale - Short Form (SCS-SF): Scale used to measure self-compassion, with higher scores reflecting greater levels of self-compassion
Change from Baseline Mindful Awareness at 2.5 Weeks, 5 Weeks, 7.5 Weeks and 11.5 | Baseline (Week 0), Pre- (Week 2.5), Mid- (Week 5), Post-Treatment (Week 7.5), and 1-month Follow-up (Week 11.5)
  Five-Facet Mindfulness Questionnaires (FFMQ): Scale used to measure mindful awareness, with higher scores reflecting greater levels of mindfulness facets

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jennine S Rawana, PhD,C.Psych., Principal Investigator — York University
Locations (1):
- York University, North York, Ontario, Canada